CLINICAL TRIAL: NCT05162014
Title: Post-authorization Safety Study (PASS) to Assess the Risk of Acute Pancreatitis in Type 2 Diabetes Mellitus (T2DM) Patients Newly Initiating Empagliflozin Compared to Other Oral Non-incretin/Non-sodium Glucose Co-transporter-2 Inhibitors (SGLT2)-Containing Glucose Lowering Drugs
Brief Title: To Assess the Risk of Acute Pancreatitis in Patients With Type 2 Diabetes Mellitus Treated With Empagliflozin
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0201
Record Dates: First submitted 2021-12-09; First posted 2021-12-17 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pooled Empagliflozin: Patients with type 2 diabetes mellitus (T2DM) and new initiators of empagliflozin on a background of metformin, between 1-Aug-2014 and the latest data-cut available in IBM MarketScan Commercial Claims and Encounters (CCAE)/ Medicare Supplemental (MDCR) 30-Sep-2020 and Optum Clinformatics® Data Mart (CDM) 31-Mar-202, who were enrolled for a minimum of 6 months in the US claims databases before index treatment initiation
  Interventions: Drug: empagliflozin
- Pooled Sulfonylureas (SUs): Patients with type 2 diabetes mellitus (T2DM) and new initiators of Sulfonylureas (SUs) on a background of metformin, between 1-Aug-2014 and the latest data-cut available in IBM MarketScan Commercial Claims and Encounters (CCAE)/ Medicare Supplemental (MDCR) 30-Sep-2020 and Optum Clinformatics® Data Mart (CDM) 31-Mar-202, who were enrolled for a minimum of 6 months in the US claims databases before index treatment initiation
  Interventions: Drug: Oral non-incretin/non-sodium glucose co-transporter-2 inhibitors (SGLT2)-containing hypoglycaemic agents

INTERVENTIONS:
Drug: empagliflozin — empagliflozin
  Groups: Pooled Empagliflozin
Drug: Oral non-incretin/non-sodium glucose co-transporter-2 inhibitors (SGLT2)-containing hypoglycaemic agents — Oral non-incretin/non-sodium glucose co-transporter-2 inhibitors (SGLT2)-containing hypoglycaemic agents
  Groups: Pooled Sulfonylureas (SUs)

SUMMARY:
To compare the risk of acute pancreatitis in patients with Type 2 diabetes mellitus (T2DM) newly initiating empagliflozin to that of patients newly initiating other oral non-incretin/non-Sodium glucose co-transporter-2 inhibitor (SGLT2i)-containing hypoglycemic agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years old
* A diagnosis of Type 2 diabetes mellitus (T2DM) as demonstrated by at least one qualifying diagnosis code from any encounter type recorded in the claims in the 6 months prior to the drug initiation.
* Patients initiating empagliflozin (as monotherapy, on a background of metformin, or on a background of metformin and Sulfonylurea (SU)) or qualifying comparator (metformin monotherapy, SU on a background of metformin, or Thiazolidinediones (TZD) on a background of metformin and SU) during the study period.
* Have at least 6 months of continuous registration in the database prior to initiation of empagliflozin or a comparator drug.

Exclusion Criteria:

* Patients with missing or ambiguous age or sex information.
* Use of a Sodium glucose co-transporter-2 inhibitor (SGLT2i), Dipeptidyl peptidase 4 inhibitors (DPP-4i) or Glucagon-like peptide-1 receptor agonist (GLP-1 RA) in the 6 months prior to study drug initiation.
* Chronic use of insulin in the outpatient setting in the 6 months prior to the study drug initiation. This criterion will help us to remove severe cases of diabetes and reduce the risk of residual confounding as diabetes is a risk factor for developing acute pancreatitis.
* Patients with type 1 diabetes mellitus (T1DM) defined as at least 1 inpatient or outpatient International Classification of Diseases Ninth Revision, Clinical Modification (ICD-9-CM) diagnosis code of 250.x1 or 250.x3 or International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) diagnosis code of E10.x in the 6 months prior to the study drug initiation.
* Patients with secondary diabetes or gestational diabetes in the 6 months prior to the study drug initiation.
* Claims for acute or chronic pancreatitis, pancreatic cancer, or other disease of the pancreas any time prior to the study drug initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a recorded diagnosis of Type 2 diabetes mellitus (T2DM) who initiated empagliflozin or other oral non-incretin/non-Sodium glucose co-transporter-2 inhibitor (SGLT2i)-containing hypoglycaemic agents (metformin, Sulfonylurea (SU), or Thiazolidinediones (TZD)) between 1 August 2014 and 31 October 2020 will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 494679 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim International GmbH, Ingelheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Post-authorization safety study based on existing data between 1-Aug-2014 and the latest data-cut available in IBM MarketScan (30-Sep-2020) and Optum Clinformatics® Data Mart (CDM) 31-Mar-2021. The study aimed to assess the risk of acute pancreatitis in type 2 diabetes mellitus (T2DM) patients newly initiated in empagliflozin to that of newly initiated in other oral non incretin/non-sodium glucose co-transporter-2 inhibitors (SGLT2i)-based glucose lowering drugs. More details in Limitations.
Pre-assignment Details: Every patient who fulfilled inclusion and exclusion criteria was selected until the required sample size was achieved.
Groups:
- Pooled Empagliflozin: Patients with type 2 diabetes mellitus (T2DM) and new initiators of empagliflozin on a background of metformin, between 1-Aug-2014 and the latest data-cut available in IBM MarketScan Commercial Claims and Encounters (CCAE)/ Medicare Supplemental (MDCR) 30-Sep-2020 and Optum Clinformatics® Data Mart (CDM) 31-Mar-2021, who were enrolled for a minimum of 6 months in the US claims databases before index treatment initiation
- Pooled Sulfonylureas (SUs): Patients with type 2 diabetes mellitus (T2DM) and new initiators of Sulfonylureas (SUs) on a background of metformin, between 1-Aug-2014 and the latest data-cut available in IBM MarketScan Commercial Claims and Encounters (CCAE)/ Medicare Supplemental (MDCR) 30-Sep-2020 and Optum Clinformatics® Data Mart (CDM) 31-Mar-2021, who were enrolled for a minimum of 6 months in the US claims databases before index treatment initiation
Period: Overall Study
Arm/Group | Pooled Empagliflozin | Pooled Sulfonylureas (SUs)
Started | 72661 | 422018
Pooled- PS Matched (Matched on propensity scores) | 72621 | 72621
Completed | 72661 | 422018
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with type 2 diabetes mellitus (T2DM) and new initiators of empagliflozin or sulfonylureas (SUs), who were enrolled between 1 August 2014 and the latest data-cut available in IBM MarketScan CCAE/MDCR (30 September 2020) and Optum CDM (31 March 2021).
Groups:
- Pooled Empagliflozin - PS Matched: Patients with type 2 diabetes mellitus (T2DM) and new initiators of empagliflozin on a background of metformin, between 1-Aug-2014 and the latest data-cut available in IBM MarketScan Commercial Claims and Encounters (CCAE)/ Medicare Supplemental (MDCR) 30-Sep-2020 and Optum Clinformatics® Data Mart (CDM) 31-Mar-2021, who were enrolled for a minimum of 6 months in the US claims databases before index treatment initiation and matched on propensity scores.
- Pooled Sulfonylureas (SUs) - PS Matched: Patients with type 2 diabetes mellitus (T2DM) and new initiators of Sulfonylureas (SUs) on a background of metformin, between 1-Aug-2014 and the latest data-cut available in IBM MarketScan Commercial Claims and Encounters (CCAE)/ Medicare Supplemental (MDCR) 30-Sep-2020 and Optum Clinformatics® Data Mart (CDM) 31-Mar-2021, who were enrolled for a minimum of 6 months in the US claims databases before index treatment initiation and matched on propensity scores
- Total: Total of all reporting groups
Arm/Group | Pooled Empagliflozin - PS Matched | Pooled Sulfonylureas (SUs) - PS Matched | Total
Number analyzed (Participants) | 72621 | 72621 | 145242
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.67 (11.53) | 56.77 (11.73) | 56.7 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30253 | 30442 | 60695
  Male | 42368 | 42179 | 84547
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Acute Pancreatitis
Description: Incidence rate of acute pancreatitis per number of person-years, defined as an acute pancreatitis diagnosis from any of the inpatient (not restricted to the primary diagnosis), outpatient, or emergency contacts diagnoses (ICD-9-CM 577.0 or ICD-10-CM K85) and a lipase measure within +/- 7 days of the acute pancreatitis diagnosis (using LOINC code of 3040-3 and 2572-6 or CPT code of 83690 for lipase) and an abdominal ultrasound (using CPT codes of 76700 and 76705) within +/- 7 days of the acute pancreatitis diagnosis. The incidence rate was reported as the number of events (counts the first event per patient) divided by the total number of person-years at risk during follow-up (1/(1000*person-years)).
Time Frame: From August 2014 to March 2021 (the study period). Up to 79 months.
Population: Pooled unmatched and 1:1 propensity scores (PS) matched cohort of patients with type 2 diabetes mellitus (T2DM) and new initiators of empagliflozin or sulfonylureas (SUs), who were enrolled between 1 August 2014 and the latest data-cut available in IBM MarketScan CCAE/MDCR (30 September 2020) and Optum CDM (31 March 2021). Primary analysis represented an 'as treated' approach.
Measure: Number (95% Confidence Interval); unit: Events per 1,000 person-years
Arm/Group | Pooled Empagliflozin - PS Matched | Pooled Sulfonylureas (SUs) - PS Matched
Number analyzed (Participants) | 72621 | 72621
Events per 1,000 person-years | 10.30 [9.29 to 11.39] | 11.65 [10.59 to 12.77]
Statistical Analysis 1: Comparison: Pooled Empagliflozin - PS Matched vs Pooled Sulfonylureas (SUs) - PS Matched; Test type: Other; Regression, Cox; Cox proportional hazards regression models based on time-to-first acute pancreatitis used to estimate the hazard ratios; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.76 to 1.02]

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: As this is a non-interventional study with secondary use of data, safety reporting on an individual case level is not applicable. All-Cause Mortality, Serious Adverse Events and Other Adverse Events were not collected in the database. "0" total Number of Participants at Risk means "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed".
Arm/Group | Pooled Empagliflozin - PS Matched | Pooled Sulfonylureas (SUs) - PS Matched
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was a Non interventional study (NIS) based on existing data. Therefore, the study might be subject to potential residual confounding due to the absence of certain key data.

In November 2021, an initial feasibility assessment was conducted which showed that the therapy cohort Empagliflozin vs. Sulfonylurea (SU) reported the highest number of empagliflozin initiators and was the only adequately powered line of therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT05162014/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT05162014/SAP_001.pdf